CLINICAL TRIAL: NCT04112186
Title: Neuroimaging Response Inhibition and Salience Attribution Changes During Mindfulness-based Treatment of Human Heroin Addiction
Brief Title: Mindfulness-Oriented Recovery Enhancement (MORE) in Heroin Addiction
Acronym: MORE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: University of Utah (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Rita Goldstein, Professor of Psychiatry and Neuroscience, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 18-0878; 1R01AT010627-01 (NIH)
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Opiate Use Disorder
Keywords: Mindfulness; Opiate Use Disorder; Drug Cue Reactivity; Inhibitory Control; Salience Attribution

STUDY DESIGN:
Intervention Model Description: Individuals with opiate use disorder (iOUD) will be randomized to one of two 8-weeks of group therapy and scanned with magnetic resonance imaging (MRI) immediately before and after treatment. Functional MRI (fMRI) scans during select tasks and at rest will assess responsiveness and connectivity of neural networks underlying impairments in Response Inhibition and Salience Attribution (iRISA). Structural MRI will assess the morphological integrity of the neural networks. A follow-up visit will take place 3 months after the second MRI scan.
  Healthy controls will be scanned at similar time intervals. Data collected from healthy control subjects will be used for comparative analyses.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The PI and the majority of study personnel, including the study statistician, will be blinded to the treatment assignment until the database is unlocked. Assessors (of endpoints) will also be blinded to treatment assignment. That is, treatment allocation will only be known by selected research associates who are not involved in assessment or treatment. The selected research associates who are unblinded will handle randomization and preparation of any unblinded reports (if required); they will not have access to the data and no involvement in data monitoring or analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral group therapy 1 (Experimental): 8-weeks of group therapy
  Interventions: Behavioral: Behavioral group therapy #1
- Behavioral group therapy 2 (Active Comparator): 8-weeks of group therapy
  Interventions: Behavioral: Behavioral group therapy #2

INTERVENTIONS:
Behavioral: Behavioral group therapy #1 — Participants will participate in an 8-weeks of group therapy that uses psychological principles including mindfulness training, and could help decrease cravings for heroin and increase general well-being.
  Arms: Behavioral group therapy 1
Behavioral: Behavioral group therapy #2 — Participants will participate in an 8-weeks of group therapy that uses psychological principles (but not including mindfulness training) and could help decrease craving for heroin and increase general well-being.
  Arms: Behavioral group therapy 2

SUMMARY:
In this study, neuroimaging of reward processing, drug cue reactivity and inhibitory control is used before and immediately after 8 weeks of two types of group therapy in individuals with opioid addiction; clinical outcomes will be assessed before, immediately and three months after treatment. Results could point to factors that track and predict recovery with treatment, offering clinicians markers that can be used for enhancing precision medicine with the goal of reducing morbidity and mortality associated with opiate addiction.

DETAILED DESCRIPTION:
Over the past 15 years, the US has been affected by increasing prescription and illicit opiate/opioid abuse, addiction, and overdose. Research into the enhancement of treatment options for individuals with opiate/opioid use disorder (iOUD) is clearly a priority. The development of neuroscience-informed behavioral therapies that could be used as adjuncts to improve effectiveness of medication-assisted interventions in iOUD is a national priority, a response to the opiate crisis. This study measures the neural correlates of cognitive function and reward processing as potentially contributing to and predictive of the impact of an 8-week group therapy on addiction outcome in iOUD. Using a pre-post randomized treatment design with a 3-months follow-up, this study will examine the impact of group therapy, as add-on to methadone maintenance, on neural functional and structural plasticity, and clinical outcomes (including daily ecological momentary assessments), in treatment-seeking iOUD (with primary use of heroin). Treatment-seeking iOUD will be randomized to 8-weeks of one of two of group therapies and scanned with magnetic resonance imaging (MRI) immediately before and after treatment. Healthy controls will be scanned at similar time intervals. Clinical outcome will be assessed during, immediately after and 3-months after therapy. Results may help identify individual variability in the brain regions/circuits that support reward processing, including cue reactivity, and inhibitory control and that could change with, and predict, response to treatment, ultimately contributing to precision medicine in OUD.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and give informed consent
* Males and Females 18-64 years of age
* DSM-5 diagnosis of OUD with heroin as the primary drug of choice
* Stabilized on methadone or other form of MAT.

Inclusion criteria for healthy controls:

- The same as inclusion criteria 1-2 above; dependence on nicotine or caffeine is non-exclusionary.

Exclusion Criteria:

* DSM-5 diagnosis for schizophrenia or developmental disorder (e.g., autism)
* Head trauma with loss of consciousness
* History of neurological disease of central origin including seizures
* Cardiovascular disease including high blood pressure and/or other medical conditions, including metabolic, endocrinological,oncological or autoimmune diseases, and infectious diseases common in iOUD including Hepatitis B and C or HIV/AIDS
* Metal implants or other MR contraindications

Exclusion criteria for healthy control subjects:

- The same, except history of any drug use disorder is prohibitive.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 157 (Actual)
Dates: Start 2020-06-21 (Actual); Primary Completion 2031-03-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in fMRI BOLD signal during tasks of reward | baseline and 3 months after enrollment
  Change in fMRI blood-oxygen-level dependent (BOLD) signal acquired during tasks of reward at the 2nd MRI conducted immediately after the 8-week group therapy (about 3 months after enrollment) as compared to baseline MRI. The reward task uses symbols of gain/win and has been shown to elicit BOLD activations in the brain's reward network.
Change in fMRI BOLD signal for control reactivity | baseline and 3 months enrollment
  Change in fMRI blood-oxygen-level dependent (BOLD) signal acquired during control reactivity at the 2nd MRI conducted immediately after the 8-week group therapy (about 3 months after enrollment) as compared to baseline MRI.
Change in fMRI BOLD signal for cue reactivity | baseline and 3 months enrollment
  Change in fMRI blood-oxygen-level dependent (BOLD) signal acquired during cue reactivity at the 2nd MRI conducted immediately after the 8-week group therapy (about 3 months after enrollment) as compared to baseline MRI.
Change in fMRI BOLD signal acquired during resting-state functional connectivity | baseline and 3 months after treatment
  Change in fMRI blood-oxygen-level dependent (BOLD) signal acquired during resting-state functional connectivity at the 2nd MRI conducted immediately after the 8-week group therapy (about 3 months after enrollment) as compared to baseline MRI. This method captures the synchronicity of low-frequency, spontaneous fluctuations in blood oxygen level-dependent signals that reflect fluctuations in neuronal activity between brain regions in the absence of external stimulation.
Change in MRI Voxel-Based Morphometry (VBM) measure | baseline and 3 months after treatment
  Change in MRI VBM measure for grey matter volume at the 2nd MRI conducted immediately after the 8-week group therapy (about 3 months after enrollment) as compared to baseline MRI. Voxel Based Morphometry is a whole-brain, fully automated, unbiased, MRI analysis technique used to detect regionally specific differences in brain tissue composition using a voxel-wise comparison across participants.
Change in Urine drug test | baseline and 3 months after treatment
  Urine drug test at 3 months after treatment as compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Rita Goldstein, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Nelly Alia-Klein, PhD, Study Director — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Relevant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal.Any purpose.Proposals should be directed to rita.goldstein@mssm.edu. To gain access, data requestors will need to sign a data access agreement.